CLINICAL TRIAL: NCT07298954
Title: Sequential Combined Versus Single-Strategy Adrenal Venous Sampling for Primary Aldosteronism: A Multicenter, Randomized Trial
Brief Title: Sequential Combined Versus Single-Strategy Adrenal Venous Sampling for Primary Aldosteronism(SCOPE)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shumin Yang (Other)
Collaborators: First Affiliated Hospital of Kunming Medical University (Other); The First Affiliated Hospital of Nanchang University (Other); The People's Hospital of Chuxiong Yi Autonomous Prefecture (Unknown)
Responsible Party: Sponsor-Investigator, Shumin Yang, Primary investigator, Chongqing Medical University
Organization: Chongqing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SCOPE PA
Record Dates: First submitted 2025-12-10; First posted 2025-12-23 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Primary Aldosteronism
Keywords: Primary Aldosteronism; Adrenal venous sampling; sequential combined AVS; non-ACTH-stimulated; ACTH-stimulated AVS; complete biochemical remission rate
MeSH Terms: conditions — Hyperaldosteronism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- sequential combined AVS (Experimental): non-ACTH-stimulated followed by ACTH-stimulated AVS
  Interventions: Diagnostic Test: sequential combined AVS
- non-ACTH-stimulated AVS (No Intervention): non-ACTH-stimulated AVS
- ACTH-stimulated AVS (No Intervention): ACTH-stimulated AVS

INTERVENTIONS:
Diagnostic Test: sequential combined AVS — non-ACTH-stimulated followed by ACTH-stimulated AVS
  Arms: sequential combined AVS

SUMMARY:
This study is a prospective, multicenter, randomized clinical trial aimed to compare the impact of three AVS diagnostic strategies on the clinical outcomes of patients with primary aldosteronism. The strategies include sequential combined AVS (non-ACTH-stimulated followed by ACTH-stimulated AVS), non- ACTH-stimulated AVS alone, and ACTH-stimulated AVS alone. The findings of this study will provide critical evidence for the clinical practice standards of AVS.

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized controlled clinical trial. This study will be led by the First Affiliated Hospital of Chongqing Medical University, with Chuxiong Yi Autonomous Prefecture People's Hospital, the First Affiliated Hospital of Kunming Medical University, and the First Affiliated Hospital of Nanchang Medical University serving as collaborating centers. According to the inclusion and exclusion criteria, eligible patients with confirmed primary aldosteronism (PA) will be enrolled and randomly assigned in a 1:1:1 ratio to one of the following groups: sequential combined AVS, non-ACTH-stimulated AVS alone, and ACTH-stimulated AVS alone. These stratifications will guide clinical treatment decisions, either surgical therapy or medical therapy, and patients will be followed to evaluate their clinical outcomes. The primary outcome is the treatment response rate at 6-month follow-up, which will be compared among the three groups.

ELIGIBILITY:
Inclusion Criteria:

* Fully understand the study process, voluntarily agree to participate, and sign informed consent.
* Diagnosed with primary aldosteronism. # Age 18-70 years with hypertension, any sex.

Exclusion Criteria:

* Patients for whom AVS can be bypassed: Typical BPA (normal serum potassium and plasma aldosterone concentration (PAC) < 110 pg/mL, eligible for direct medical therapy); Typical UPA (PAC ≥ 200 pg/mL, plasma renin concentration (PRC) ≤ 5 μIU/mL, spontaneous hypokalemia, unilateral adrenal adenoma ≥ 1 cm with normal contralateral adrenal on CT or 68Ga-Pentixafor PET-CT indicating unilateral functional tumor, eligible for direct surgery);
* Refusal of AVS or surgery, or contraindication to surgery.
* Allergy to ACTH or contrast agents.
* Combined with autonomous cortisol secretion (1 mg overnight dexamethasone suppression test cortisol ≥ 50 nmol/L).
* Early-onset hypertension (<20 years) with hypokalemia and family history, suggestive of familial hyperaldosteronism or Liddle syndrome.
* Imaging cannot exclude pheochromocytoma or adrenocortical carcinoma (nodule ≥ 4 cm, CT ≥ 20 HU, or MRI suggestive).
* Active malignancy.
* Previous adrenal surgery.
* Chronic glucocorticoid use that cannot be discontinued.
* Adrenal insufficiency requiring hormone replacement.
* Pregnancy or breastfeeding; history of alcohol or substance abuse, or inability to cooperate due to psychiatric disorders.
* NYHA class III-IV heart failure or hospitalization for worsening heart failure in the past 3 months, stroke or acute coronary syndrome in past 3 months, severe anemia (Hb < 60 g/L), severe liver or renal disease (ALT ≥ 3×upper limit; eGFR <30 mL/min/1.73 m2 or dialysis), systemic inflammatory response syndrome (SIRS), poorly controlled diabetes (FBG ≥ 13.3 mmol/L), severe obesity (BMI ≥ 35 kg/m2), untreated aneurysm, or other conditions severely interfering with study participation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 456 (Estimated)
Dates: Start 2025-12-25 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of complete biochemical remission | At 6 months of follow-up
  Blood was drawn to measure aldosterone, renin and potassium.According to PASO criteria, outcomes of adrenalectomy for unilateral primary aldosteronism were classified into complete, partial, and absent success, for both clinical and biochemical outcomes.The proportion of complete biochemical remission according to PASO consensus criteria.

SECONDARY OUTCOMES:
The proportion of complete clinical remission | At 6 months of follow-up
  Blood was drawn to measure aldosterone, renin and potassium.According to PASO criteria, outcomes of adrenalectomy for unilateral primary aldosteronism were classified into complete, partial, and absent success, for both clinical and biochemical outcomes.The proportion of complete clinical remission according to PASO consensus criteria.
The proportion of complete biochemical response rate | At 6 months of follow-up
  Blood was drawn to measure aldosterone, renin and potassium.According to PAMO criteria, outcomes of medication for bilateral primary aldosteronism were classified into complete, partial, and absent response, for both clinical and biochemical outcomes.The proportion of complete biochemical response according to PAMO consensus criteria.
The proportion of complete clinical response rate | At 6 months of follow-up
  Blood was drawn to measure aldosterone, renin and potassium.According to PAMO criteria, outcomes of medication for bilateral primary aldosteronism were classified into complete, partial, and absent response, for both clinical and biochemical outcomes.The proportion of complete clinical response according to PAMO consensus criteria.
Comparison of adverse events | At 6 months of follow-up
  The occurrence of adverse events was recorded, including adrenal vein rupture, peripheral puncture site complications including femoral vein thrombosis, puncture site hematoma, ACTH allergy, and anaphylactic shock., etc.
In surgical population, the proportion of complete biochemical remission | At 6 months of follow-up
  Blood was drawn to measure aldosterone, renin and potassium.According to PASO criteria, outcomes of adrenalectomy for unilateral primary aldosteronism were classified into complete, partial, and absent success, for both clinical and biochemical outcomes.The proportion of complete biochemical remission according to PASO consensus criteria.
In surgical population, the proportion of complete clinical remission | At 6 months of follow-up
  Blood was drawn to measure aldosterone, renin and potassium.According to PASO criteria, outcomes of adrenalectomy for unilateral primary aldosteronism were classified into complete, partial, and absent success, for both clinical and biochemical outcomes.The proportion of complete clinical remission according to PASO consensus criteria.
In medication population, the proportion of complete biochemical response rate | At 6 months of follow-up
  Blood was drawn to measure aldosterone, renin and potassium.According to PAMO criteria, outcomes of medication for bilateral primary aldosteronism were classified into complete, partial, and absent response, for both clinical and biochemical outcomes.The proportion of complete biochemical response according to PAMO consensus criteria.
In medication population, the proportion of complete clinical response rate | At 6 months of follow-up
  Blood was drawn to measure aldosterone, renin and potassium.According to PAMO criteria, outcomes of medication for bilateral primary aldosteronism were classified into complete, partial, and absent response, for both clinical and biochemical outcomes.The proportion of complete clinical response according to PAMO consensus criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Shumin Yang, Study Chair — the Chongqing Primary Aldosteronism Study (CONPASS) Group
Locations (1):
- The First Affilated Hospital of Chongqing Medical University, Chongqing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Monticone S, Burrello J, Tizzani D, Bertello C, Viola A, Buffolo F, Gabetti L, Mengozzi G, Williams TA, Rabbia F, Veglio F, Mulatero P. Prevalence and Clinical Manifestations of Primary Aldosteronism Encountered in Primary Care Practice. J Am Coll Cardiol. 2017 Apr 11;69(14):1811-1820. doi: 10.1016/j.jacc.2017.01.052. PMID 28385310
- [Result] Rossi GP, Bernini G, Caliumi C, Desideri G, Fabris B, Ferri C, Ganzaroli C, Giacchetti G, Letizia C, Maccario M, Mallamaci F, Mannelli M, Mattarello MJ, Moretti A, Palumbo G, Parenti G, Porteri E, Semplicini A, Rizzoni D, Rossi E, Boscaro M, Pessina AC, Mantero F; PAPY Study Investigators. A prospective study of the prevalence of primary aldosteronism in 1,125 hypertensive patients. J Am Coll Cardiol. 2006 Dec 5;48(11):2293-300. doi: 10.1016/j.jacc.2006.07.059. Epub 2006 Nov 13. PMID 17161262
- [Result] Xu Z, Yang J, Hu J, Song Y, He W, Luo T, Cheng Q, Ma L, Luo R, Fuller PJ, Cai J, Li Q, Yang S; Chongqing Primary Aldosteronism Study (CONPASS) Group. Primary Aldosteronism in Patients in China With Recently Detected Hypertension. J Am Coll Cardiol. 2020 Apr 28;75(16):1913-1922. doi: 10.1016/j.jacc.2020.02.052. PMID 32327102
- [Result] Libianto R, Russell GM, Stowasser M, Gwini SM, Nuttall P, Shen J, Young MJ, Fuller PJ, Yang J. Detecting primary aldosteronism in Australian primary care: a prospective study. Med J Aust. 2022 May 2;216(8):408-412. doi: 10.5694/mja2.51438. Epub 2022 Feb 25. PMID 35218017
- [Result] Mulatero P, Sechi LA, Williams TA, Lenders JWM, Reincke M, Satoh F, Januszewicz A, Naruse M, Doumas M, Veglio F, Wu VC, Widimsky J. Subtype diagnosis, treatment, complications and outcomes of primary aldosteronism and future direction of research: a position statement and consensus of the Working Group on Endocrine Hypertension of the European Society of Hypertension. J Hypertens. 2020 Oct;38(10):1929-1936. doi: 10.1097/HJH.0000000000002520. PMID 32890265
- [Result] Hundemer GL, Curhan GC, Yozamp N, Wang M, Vaidya A. Renal Outcomes in Medically and Surgically Treated Primary Aldosteronism. Hypertension. 2018 Sep;72(3):658-666. doi: 10.1161/HYPERTENSIONAHA.118.11568. PMID 29987110
- [Result] Funder JW, Carey RM, Mantero F, Murad MH, Reincke M, Shibata H, Stowasser M, Young WF Jr. The Management of Primary Aldosteronism: Case Detection, Diagnosis, and Treatment: An Endocrine Society Clinical Practice Guideline. J Clin Endocrinol Metab. 2016 May;101(5):1889-916. doi: 10.1210/jc.2015-4061. Epub 2016 Mar 2. PMID 26934393
- [Result] Song Y, Yang J, Shen H, Ng E, Fuller PJ, Feng Z, Hu J, Ma L, Yang Y, Du Z, Wang Y, Luo T, He W, Li Q, Wu FF, Yang S; represent for the Chongqing Primary Aldosteronism Study (CONPASS) Group. Development and validation of model for sparing adrenal venous sampling in diagnosing unilateral primary aldosteronism. J Hypertens. 2022 Sep 1;40(9):1692-1701. doi: 10.1097/HJH.0000000000003197. Epub 2022 Jul 22. PMID 35881462
- [Result] Adler GK, Stowasser M, Correa RR, Khan N, Kline G, McGowan MJ, Mulatero P, Murad MH, Touyz RM, Vaidya A, Williams TA, Yang J, Young WF, Zennaro MC, Brito JP. Primary Aldosteronism: An Endocrine Society Clinical Practice Guideline. J Clin Endocrinol Metab. 2025 Aug 7;110(9):2453-2495. doi: 10.1210/clinem/dgaf284. PMID 40658480
- [Result] Chee NYN, Abdul-Wahab A, Libianto R, Gwini SM, Doery JCG, Choy KW, Chong W, Lau KK, Lam Q, MacIsaac RJ, Chiang C, Shen J, Young MJ, Fuller PJ, Yang J. Utility of adrenocorticotropic hormone in adrenal vein sampling despite the occurrence of discordant lateralization. Clin Endocrinol (Oxf). 2020 Oct;93(4):394-403. doi: 10.1111/cen.14220. Epub 2020 Jun 15. PMID 32403203
- [Result] Elliott P, Holmes DT. Adrenal vein sampling: substantial need for technical improvement at regional referral centres. Clin Biochem. 2013 Oct;46(15):1399-404. doi: 10.1016/j.clinbiochem.2013.04.004. Epub 2013 Apr 16. PMID 23603377
- [Result] Laurent I, Astere M, Zheng F, Chen X, Yang J, Cheng Q, Li Q. Adrenal venous sampling with or without adrenocorticotropic hormone stimulation: A meta-analysis. J Clin Endocrinol Metab. 2018 Nov 6. doi: 10.1210/jc.2018-01324. Online ahead of print. PMID 30403797
- [Result] Monticone S, Satoh F, Giacchetti G, Viola A, Morimoto R, Kudo M, Iwakura Y, Ono Y, Turchi F, Paci E, Veglio F, Boscaro M, Rainey W, Ito S, Mulatero P. Effect of adrenocorticotropic hormone stimulation during adrenal vein sampling in primary aldosteronism. Hypertension. 2012 Apr;59(4):840-6. doi: 10.1161/HYPERTENSIONAHA.111.189548. Epub 2012 Feb 13. PMID 22331382
- [Result] Rossi GP, Pitter G, Bernante P, Motta R, Feltrin G, Miotto D. Adrenal vein sampling for primary aldosteronism: the assessment of selectivity and lateralization of aldosterone excess baseline and after adrenocorticotropic hormone (ACTH) stimulation. J Hypertens. 2008 May;26(5):989-97. doi: 10.1097/HJH.0b013e3282f9e66a. PMID 18398342
- [Result] Rossi GP, Ganzaroli C, Miotto D, De Toni R, Palumbo G, Feltrin GP, Mantero F, Pessina AC. Dynamic testing with high-dose adrenocorticotrophic hormone does not improve lateralization of aldosterone oversecretion in primary aldosteronism patients. J Hypertens. 2006 Feb;24(2):371-9. doi: 10.1097/01.hjh.0000202818.10459.96. PMID 16508586
- [Result] Seccia TM, Miotto D, De Toni R, Pitter G, Mantero F, Pessina AC, Rossi GP. Adrenocorticotropic hormone stimulation during adrenal vein sampling for identifying surgically curable subtypes of primary aldosteronism: comparison of 3 different protocols. Hypertension. 2009 May;53(5):761-6. doi: 10.1161/HYPERTENSIONAHA.108.128553. Epub 2009 Apr 6. PMID 19349554
- [Result] Rossitto G, Amar L, Azizi M, Riester A, Reincke M, Degenhart C, Widimsky J, Naruse M, Deinum J, Schultzekool L, Kocjan T, Negro A, Rossi E, Kline G, Tanabe A, Satoh F, Rump LC, Vonend O, Willenberg HS, Fuller P, Yang J, Nian Chee NY, Magill SB, Shafigullina Z, Quinkler M, Oliveras A, Chang CC, Wu VC, Somloova Z, Maiolino G, Barbiero G, Battistel M, Lenzini L, Quaia E, Pessina AC, Rossi GP. Subtyping of Primary Aldosteronism in the AVIS-2 Study: Assessment of Selectivity and Lateralization. J Clin Endocrinol Metab. 2020 Jun 1;105(6):dgz017. doi: 10.1210/clinem/dgz017. PMID 31536622
- [Result] Takeda Y, Umakoshi H, Takeda Y, Yoneda T, Kurihara I, Katabami T, Ichijo T, Wada N, Yoshimoto T, Ogawa Y, Kawashima J, Sone M, Takahashi K, Watanabe M, Matsuda Y, Kobayashi H, Shibata H, Kamemura K, Otsuki M, Fujii Y, Yamamto K, Ogo A, Yanase T, Suzuki T, Naruse M; JPAS Study Group. Impact of adrenocorticotropic hormone stimulation during adrenal venous sampling on outcomes of primary aldosteronism. J Hypertens. 2019 May;37(5):1077-1082. doi: 10.1097/HJH.0000000000001964. PMID 30601318
- [Result] Yatabe M, Bokuda K, Yamashita K, Morimoto S, Yatabe J, Seki Y, Watanabe D, Morita S, Sakai S, Ichihara A. Cosyntropin stimulation in adrenal vein sampling improves the judgment of successful adrenal vein catheterization and outcome prediction for primary aldosteronism. Hypertens Res. 2020 Oct;43(10):1105-1112. doi: 10.1038/s41440-020-0445-x. Epub 2020 Apr 30. PMID 32355223
- [Result] Yozamp N, Hundemer GL, Moussa M, Underhill J, Fudim T, Sacks B, Vaidya A. Adrenocorticotropic Hormone-Stimulated Adrenal Venous Sampling Underestimates Surgically Curable Primary Aldosteronism: A Retrospective Cohort Study and Review of Contemporary Studies. Hypertension. 2021 Jul;78(1):94-103. doi: 10.1161/HYPERTENSIONAHA.121.17248. Epub 2021 May 17. PMID 33993726
- [Result] Yang S, Du Z, Zhang X, Zhen Q, Shu X, Yang J, Song Y, Yang Y, Li Q, Hu J; Chongqing Primary Aldosteronism Study (CONPASS) Group. Corticotropin Stimulation in Adrenal Venous Sampling for Patients With Primary Aldosteronism: The ADOPA Randomized Clinical Trial. JAMA Netw Open. 2023 Oct 2;6(10):e2338209. doi: 10.1001/jamanetworkopen.2023.38209. PMID 37870836
- [Result] Preston CA, Yong EXZ, Marginson B, Farrell SG, Sawyer MP, Hashimura H, Derbyshire MM, MacIsaac RJ, Sachithanandan N. Utility of Adrenal Vein Sampling With and Without Ultra-Low Dose ACTH Infusion in the Diagnostic Evaluation of Primary Aldosteronism. Endocrinol Diabetes Metab. 2024 Sep;7(5):e70001. doi: 10.1002/edm2.70001. PMID 39207956
- [Result] Hu J, Xu T, Shen H, Song Y, Yang J, Zhang A, Ding H, Xing N, Li Z, Qiu L, Ma L, Yang Y, Feng Z, Du Z, He W, Sun Y, Cai J, Li Q, Chen Y, Yang S; Chongqing Primary Aldosteronism Study (CONPASS) Group. Accuracy of Gallium-68 Pentixafor Positron Emission Tomography-Computed Tomography for Subtyping Diagnosis of Primary Aldosteronism. JAMA Netw Open. 2023 Feb 1;6(2):e2255609. doi: 10.1001/jamanetworkopen.2022.55609. PMID 36795418
- [Result] Williams TA, Lenders JWM, Mulatero P, Burrello J, Rottenkolber M, Adolf C, Satoh F, Amar L, Quinkler M, Deinum J, Beuschlein F, Kitamoto KK, Pham U, Morimoto R, Umakoshi H, Prejbisz A, Kocjan T, Naruse M, Stowasser M, Nishikawa T, Young WF Jr, Gomez-Sanchez CE, Funder JW, Reincke M; Primary Aldosteronism Surgery Outcome (PASO) investigators. Outcomes after adrenalectomy for unilateral primary aldosteronism: an international consensus on outcome measures and analysis of remission rates in an international cohort. Lancet Diabetes Endocrinol. 2017 Sep;5(9):689-699. doi: 10.1016/S2213-8587(17)30135-3. Epub 2017 May 30. PMID 28576687
- [Result] Yang J, Burrello J, Goi J, Reincke M, Adolf C, Asbach E, Brudgam D, Li Q, Song Y, Hu J, Yang S, Satoh F, Ono Y, Libianto R, Stowasser M, Li N, Zhu Q, Hong N, Nayak D, Puar TH, Wu VC, Vaidya A, Araujo-Castro M, Kocjan T, O'Toole SM, Hundemer GL, Ragnarsson O, Lacroix A, Larose S, Nakai K, Nishikawa T, Ladygina D, Turcu AF, Sholinyan J, Fardella CE, Uslar T, Quinkler M, Mulatero P, Pintus G, Rossi GP, Hahner S, Amar L, Drake WM, Varsani C, Brown MJ, Wu X, Deinum J, Freel EM, Kline G, Naruse M, Prejbisz A, Young WF Jr, Williams TA, Fuller PJ. Outcomes after medical treatment for primary aldosteronism: an international consensus and analysis of treatment response in an international cohort. Lancet Diabetes Endocrinol. 2025 Feb;13(2):119-133. doi: 10.1016/S2213-8587(24)00308-5. Epub 2025 Jan 14. PMID 39824204